CLINICAL TRIAL: NCT06544200
Title: Intra-operative Air Leak Management After Minimally Invasive Lung Segmental Resection: Randomized Comparison Between Polymeric Hydrogel Matrix and Standard of Care
Brief Title: Intra-operative Air Leak Management After Minimally Invasive Lung Segmental Resection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Padova (Other)
Responsible Party: Principal Investigator, Giovanni Maria Comacchio, Thoracic Surgeon, University Hospital Padova
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 513n/AO24
Record Dates: First submitted 2024-07-30; First posted 2024-08-09 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Lung Cancer Stage I; Lung; Node; Air Leak From Lung
Keywords: thoracoscopic surgery; Segmentectomy; Air Leak; Hydrogel Matrix
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Polymeric Hydrogel Matrix (Experimental): single application of Polymeric Hydrogel Matrix at the completion of lung resection, in patients with moderate intraoperative alveolar air leaks (30-60 ml/respiratory act), measured at the Ventilation Mechanical Test, which consists in 1 minute volumetric ventilation with a constant flow and a peak pressure of 22 cmH2O, 12 respiratory rates per minute and a positive end-expiratory pressure (PEEP) of 5 cmH2O.
  Interventions: Device: Polymeric Hydrogel Matrix
- Control Group (No Intervention): no further treatment at the completion of lung resection, in patients with moderate intraoperative alveolar air leaks (30-60 ml/respiratory act), measured at the Ventilation Mechanical Test, which consists in 1 minute volumetric ventilation with a constant flow and a peak pressure of 22 cmH2O, 12 respiratory rates per minute and a positive end-expiratory pressure (PEEP) of 5 cmH2O.

INTERVENTIONS:
Device: Polymeric Hydrogel Matrix — application of Polymeric Hydrogel Matrix along the suture line at the completion of lung resection
  Arms: Polymeric Hydrogel Matrix

SUMMARY:
In patients undergoing minimally invasive thoracoscopic surgery (video-assisted thoracoscopic surgery, or VATS), a still unsolved issue is represented by intraoperative alveolar air leaks (IOAALs), which if prolonged beyond the fifth postoperative day can lead to higher risk of complications and higher medical costs. The polymeric hydrogel matrix (PHM) is a novel tool to manage intraoperative IOAALs. The primary end-point of our study was to verify whether PHM would be able to reduce postoperative air leaks; secondary end-points were the possible reduction of the permanence time of the chest drain (CD) and the hospital length (HL) in the PHM group compared with no treatment.

DETAILED DESCRIPTION:
The management of postoperative air leaks remains an unresolved issue in pulmonary resections. This complication can be present in up to 75% of patients undergoing major lung resections; however, it often resolves spontaneously. In 8% of cases, air leaks can persist for up to 5-7 days post-surgery, and are associated with a higher risk of complications, such as prolonged chest tube duration, increased incidence of postoperative infections and higher medical and non-medical costs. Sealants are non-invasive medical devices that help reduce or eliminate air leaks and bleeding. A recent study showed an increased risk of air leaks in patients undergoing segmentectomies compared to lobar resections; this study is designed to evaluate the efficacy of intraoperative use of Polymeric Hydrogel matrix in achieving aerostasis during anatomical segmental pulmonary resections via VATS or RATS, compared to patients receiving standard of care. All patients meet the eligibility criteria and successfully undergo a minimally invasive segmentectomy will undergo intraoperative evaluation of alveolar air leaks. Those with moderate air leaks (30-60 ml/respiratory act, measured at the Ventilation Mechanical Test, which consists in 1 minute volumetric ventilation with a constant flow and a peak pressure of 22 cmH2O, 12 respiratory rates per minute and a positive end-expiratory pressure (PEEP) of 5 cmH2O), will be randomized to receive Polymeric Hydrogel matrix or no further treatment.The primary endpoint is to evaluate the efficacy in reducing postoperative air leaks secondary to the intraoperative application of Polymeric Hydrogel matrix (measured in days from the first postoperative day to the last day the air leaks are detected), compared to a control group receiving standard of care.The secondary endpoints include the evaluation of the postoperative permanence of chest tube, total length of hospital stay, medical and non-medical costs and postoperative complications up to 40 days of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* patients aged > 18 years
* undergoing anatomical pulmonary resection (segmentectomy) via VATS or RATS
* benign and/or malignant lung disease
* No known allergy to any of the components of the device

Exclusion Criteria:

* Refusal or inability to give informed consent to the study protocol
* Age < 18 years
* Pregnancy
* Chronic Kidney Failure
* Allergies or contraindications to any of the Polymeric Hydrogel Matrix components
* Patients undergoing pulmonary resections different than segmentectomy (wedge, lobectomy, bilobectomy, pneumonectomy)
* Patients undergoing open surgery
* More than one chest tube after lung resection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2023-07-15 (Actual); Primary Completion 2024-07-13 (Actual); Study Completion 2024-07-13 (Actual)

PRIMARY OUTCOMES:
presence of postoperative air leaks | days from end of surgery up to 40 days of postoperative follow-up
  The presence of postoperative air leaks from pleural drainage, from the end of surgery to the last day the air leaks are detected.

SECONDARY OUTCOMES:
Chest drain length of stay | days from the first postoperative day up to 40 days of postoperative follow-up
  The duration of pleural drainage placement from the first postoperative day until the day of its removal
In-Hospital length of stay | days from the first postoperative day up to 40 days of postoperative follow-up
  The length of hospital stay, measured from the first postoperative day until the patient is discharged from the hospital ward
Incidence of postoperative complications | days from the first postoperative day up to 40 days of postoperative follow-up
  Any complications arising in patients are recorded and assigned a severity grade according to the Clavien-Dindo classification.

CONTACTS AND LOCATIONS:
Overall Officials: Samuele Nicotra, MDF, Principal Investigator — Thoracic Surgery Unit, University Hospital of Padua
Locations (1):
- Thoracic Surgery Unit, Padua, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fuller C. Reduction of intraoperative air leaks with Progel in pulmonary resection: a comprehensive review. J Cardiothorac Surg. 2013 Apr 16;8:90. doi: 10.1186/1749-8090-8-90. PMID 23590942
- [Background] Zaraca F, Vaccarili M, Zaccagna G, Maniscalco P, Dolci G, Feil B, Perkmann R, Bertolaccini L, Crisci R. Cost-effectiveness analysis of sealant impact in management of moderate intraoperative alveolar air leaks during video-assisted thoracoscopic surgery lobectomy: a multicentre randomised controlled trial. J Thorac Dis. 2017 Dec;9(12):5230-5238. doi: 10.21037/jtd.2017.11.109. PMID 29312730
- [Background] Suzuki K, Saji H, Aokage K, Watanabe SI, Okada M, Mizusawa J, Nakajima R, Tsuboi M, Nakamura S, Nakamura K, Mitsudomi T, Asamura H; West Japan Oncology Group; Japan Clinical Oncology Group. Comparison of pulmonary segmentectomy and lobectomy: Safety results of a randomized trial. J Thorac Cardiovasc Surg. 2019 Sep;158(3):895-907. doi: 10.1016/j.jtcvs.2019.03.090. Epub 2019 Apr 9. PMID 31078312
- [Derived] Nicotra S, Comacchio GM, Mammana M, Sambataro V, Pagliarini G, Bonis A, Boemo D, Bovo P, Rebusso A, Schiavon M, Cannone G, Faccioli E, Dell'Amore A, Rea F. Air leaks management using polymeric hydrogel matrix after thoracoscopic lung segmentectomy: a single-center prospective randomized trial with a cost-effective analysis. Updates Surg. 2025 Jun 21. doi: 10.1007/s13304-025-02291-1. Online ahead of print. PMID 40543008